CLINICAL TRIAL: NCT03693248
Title: Multi-center, Randomized Controlled, Phase III Trials to Evaluate the Safety and Effectiveness After Cycles Reduction of Neoadjuvant Chemotherapy for Advanced Epithelial Ovarian, Fallopian and Primary Peritoneal Cancer
Brief Title: Reduction Of Cycles of neOadjuvant Chemotherapy for Advanced Epithelial Ovarian, Fallopian and Primary Peritoneal Cancer
Acronym: ROCOCO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0228
Record Dates: First submitted 2018-07-13; First posted 2018-10-02 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IV; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: advanced ovarian cancer; advanced fallopian cancer; advanced peritoneal cancer; neoadjuvant chemotherapy; cycles of chemotherapy; survival
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Comparison of clinical outcomes between two and three cycles of neoadjuvant chemotherapy followed by interval debulking surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two cycles of neoadjuvant chemotherapy (Experimental): * Paclitaxel (175mg/m2) and carboplatin (AUC 5.0 or 6.0) IV, D1, every three weeks.
  * Two cycles of neoadjuvant chemotherapy and four cycles of adjuvant chemotherapy.
  Interventions: Drug: Two cycles of neoadjuvant chemotherapy
- Three cycles of neoadjuvant chemotherapy (No Intervention): * Paclitaxel (175mg/m2) and carboplatin (AUC 5.0 or 6.0) IV, D1, every three weeks.
  * Three cycles of neoadjuvant chemotherapy and three cycles of adjuvant chemotherapy.

INTERVENTIONS:
Drug: Two cycles of neoadjuvant chemotherapy — Two and three cycles of neoadjuvant chemotherapy will be administered in experimental and control groups, respectively
  Other Names: paclitaxel and carboplatin
  Arms: Two cycles of neoadjuvant chemotherapy

SUMMARY:
Te hypothesized that two cycles of neoadjuvant chemotherapy followed by interval debulking surgery would improve survival in advanced epithelial ovarian, fallopian, and primary peritoneal cancer because reduction of one cycle of chemotherapy can lead to the removal of more tumor burden, compared with three cycles of neoadjuvant chemotherapy.

So the investigators aim to compare survival, rate of successful optimal cytoreductive surgery, post-operative complications, and quality of life between two and three cycles of neoadjuvant chemotherapy followed by interval debulking surgery for advanced epithelial ovarian, fallopian, and primary peritoneal cancer.

DETAILED DESCRIPTION:
Primary debulking surgery (PDS) followed by adjuvant chemotherapy is the standard treatment for advanced epithelial ovarian, fallopian and primary peritoneal cancer. However, three or four cycles of neoadjuvant chemotherapy (NAC) followed by interval debulking surgery (IDS) has been introduced in clinical setting because four randomized controlled trials related have shown a lower rate of complications in NAC followed by IDS despite the similar efficacy between PDS and NAC followed by IDS in advanced epithelial ovarian, fallopian and primary peritoneal cancers. However, these trials have some limitations that the rate of optimal cytoreduction defined as the size of residual tumor <1 cm was about 40%, which was a disappointed result not showing the surgical effect improving survival. Nevertheless, more treatment strategies using NAC followed by IDS should be investigated because NAC followed by IDS has been already known as another standard treatment due to the safety.

A recent meta-analysis has reported that reduction of one cycle of neoadjuvant chemotherapy may increase overall survival of 4.1 months because it can induce surgical resection of more visible tumors with drug-resistant. Moreover, a related clinical trial has shown that hyperthermic intraperitoneal chemotherapy (HIPEC) may increase survival in patients with advanced ovarian cancer who received three cycles of neoadjuvant chemotherapy because HIPEC can kill drug-resistant invisible tumor cells which were not resected during IDS. Thus, the investigators designed a phase 3, multicenter, randomized controlled trial for comparing survival, clinical outcomes and quality of life between two and three cycles of NAC followed by IDS, and thereby will investigate the efficacy and safety of reduction of one cycle of NAC.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-80 years old
2. Advanced epithelial ovarian, fallopian or primary peritoneal cancer diagnosed with the following methods

   * Histologic confirmation by diagnostic laparoscopic or laparotomy ② Histologic malignancy originated from female genital tract on fine needle aspiration if histological confirmation is difficult or cytologic confirmation of adenocarcinoma in ascites if fine needle aspiration is difficult, meeting the following criteria

     * Existence of the pelvic or ovarian mass
     * Identification of tumor >2 cm beyond the pelvis on CT, malignant pleural effusion by thoracentesis, extraperitoneal lymph node metastasis (cardio-phrenic, internal mammary, mediastinal, para-tracheal, supraclavicular lymph nodes or inguinal lymph nodes)
     * Cancer antigen 125 (CA-125, kU/L)/carcinoembryonic antigen (CEA, ng/ml) >25
     * if CA-125 (kU/L)/CEA (ng/ml) is 25 or less, no primary lesion on colonoscopy, gastroscopy and mammography within six weeks before randomization.
3. International Federation of Gynecology and Obstetrics (FIGO) stage IIIC to IVB disease
4. World Health Organization performance status 0-2
5. The following criteria should be met if synchronous or metachronous tumors exists.

   ① Complete remission of metachronous malignancy for at least 5 years

   ② Follicular or papillary thyroid cancer treated completely with only surgery as a synchronous tumor

   ③ Early gastric or colon cancer treated completely with only endoscopic mucosal resection as a synchronous tumor
6. Normal hematologic, renal and liver function with the following criteria White blood cell (WBC) ≥3,000/ul Absolute neutrophil count (ANC) ≥1,500/ul Platelet ≥100×103/ul Aspartate aminotransferase (AST) ≤100 IU/L Alanine aminotransferase (ALT) ≤100 IU/L Serum total bilirubin ≤1.5 mg/dL Serum creatinine ≤1.5 mg/dL
7. Absence of psychological, and socioeconomic limitations affecting participation to this trial
8. Informed consent

Exclusion Criteria:

1. Diagnosis of metachronous malignancy within five years before enrollment
2. Synchronous tumors except follicular or papillary thyroid cancer treated completely with only surgery and early gastric or colon cancer treated completely with only endoscopic mucosal resection
3. Carcinoma in situ, non-epithelial, or borderline tumor in ovary, fallopian tube, and peritoneum
4. Pregnancy
5. Medical conditions (hypertension, diabetes mellitus, infectious or cardiac disease etc.) influencing on survival
6. Clinical evidence of brain or leptomeningeal metastasis, bone metastasis
7. Other treatments affecting clinical outcomes during participation to this trial (hyperthermic intraperitoneal chemotherapy, onco-thermia, herbal medicine, etc.)
8. No informed consent

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death (by any cause, in the absence of disease progression) whichever came first, assessed up to 60 months
  the time interval from randomization date to disease recurrence or progression date

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until death due to any cause, assessed up to 60 months
  the time interval from randomization date to death or end of study date
Time to progression | From date of randomization until the date of first documented progression in the absence of death by any cause, assessed up to 60 months
  the time interval from randomization date to disease recurrence or progression except death date
Tumor response 1 | 3 weeks after completion of neoadjuvant chemotherapy, up to 6 weeks
  Tumor response after neoadjuvant chemotherapy
Tumor response 2 | 3 weeks after completion of interval debulking surgery, up to 6 weeks
  Surgical response after interval debulking surgery
Tumor response 3 | 3 weeks after completion of adjuvant chemotherapy, up to 6 weeks
  Tumor response after adjuvant chemotherapy
Radiologic evaluation of residual tumor | 3 weeks after interval debulking surgery, up to 6 weeks
  Size of post operative residual tumor on computed tomography (CT) after interval debulking surgery
Functional assessment of residual tumor | 3 weeks after neoadjuvant chemotherapy, up to 6 weeks
  Standardized uptake positron emission tomography (PET) CT
Assessment of quality of life1 | From the date of screening to the date before treatment start, 3 weeks after interval debulking surgery within 6 weeks, 3 weeks after completion of adjuvant chemotherapy up to 6 weeks, on date of visit at 6 months after completion of primary treatment
  Scoring of quality of life assessment using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Assessment of quality of life2 | From the date of screening to the date before treatment start, 3 weeks after interval debulking surgery within 6 weeks, 3 weeks after completion of adjuvant chemotherapy up to 6 weeks, on date of visit at 6 months after completion of primary treatment
  Scoring of quality of life assessment using the EORTC ovarian cancer module (EORTC QLQ-Ov28)
Assessment of quality of life3 | From the date of screening to the date before treatment start, 3 weeks after interval debulking surgery within 6 weeks, 3 weeks after completion of adjuvant chemotherapy up to 6 weeks, on date of visit at 6 months after completion of primary treatment
  Scoring of quality of life assessment using the Functional Assessment of Cancer Therapy (FACT-O)
Assessment of quality of life4 | From the date of screening to the date before treatment start, 3 weeks after interval debulking surgery within 6 weeks, 3 weeks after completion of adjuvant chemotherapy up to 6 weeks, on date of visit at 6 months after completion of primary treatment
  Scoring of quality of life assessment using the EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
Adverse events | From the date of first day of chemotherapy to the day before starting next cycle. Each cycle is 21 days.
  Evaluation of chemotherapy induced toxicity
Success rate of optimal cytoreduction | On the date of completion of interval debulking surgery, up to 24 hours
  Evaluation of optimal cytoreduction and extent of resection based on modified Korean Gynecologic Oncology Group (KGOG) operation record form and tumor burden index
Surgical complexity score (SCS) | On the date of completion of interval debulking surgery, up to 24 hours
  Evaluation of difficulty of surgical skills based on surgical complexity score Minimal 0 to maxial 18 point. Each surgery will classified into low (point ≤3), intermediate (4-7), high (≥8) Higher value means more complex surgery.
Postoperative complications 1 | Early complications: after interval debulking surgery, up to 30 days
  Incidence of early complications, and severity of complications based on Memorial Sloan Kettering Cancer Center Surgical Secondary Events Grading System
Postoperative complications 2 | Late complications: 31 days after interval debulking surgery through study completion, an average of 1 year
  Incidence of late complications, and severity of complications based on Memorial Sloan Kettering Cancer Center Surgical Secondary Events Grading System
Estimated blood loss | after interval debulking surgery up to 3 months
  Estimated blood loss (ml) based on Modified KGOG Operation Record Form
Operation time | after interval debulking surgery up to 3 months
  Operation time (min) based on Modified KGOG Operation Record Form
Transfusion | after interval debulking surgery up to 3 months
  Transfusion (count by volume of transfused RBC) based on Modified KGOG Operation Record Form
days of hospitalization | after interval debulking surgery up to 3 months
  days of hospitalization based on Modified KGOG Operation Record Form
days of management in intensive care unit | after interval debulking surgery up to 3 months
  days of management in intensive care unit based on Modified KGOG Operation Record Form

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park SJ, Shim SH, Ji YI, Kwon SH, Lee EJ, Lee M, Chang SJ, Park S, Kim SY, Lee SJ, Kim JW, Roh JW, Lee SH, Song T, Kim HS. Reduction of cycles of neoadjuvant chemotherapy for advanced epithelial ovarian, fallopian or primary peritoneal cancer (ROCOCO): study protocol for a phase III randomized controlled trial. BMC Cancer. 2020 May 6;20(1):385. doi: 10.1186/s12885-020-06886-2. PMID 32375688